CLINICAL TRIAL: NCT01061021
Title: HIV Treatment Adherence/Risk Reduction Integrated
Brief Title: HIV Prevention Intervention for People Living With HIV/AIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Seth C. Kalichman / Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H06-113; R01MH071164-04 (NIH)
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infections
Keywords: HIV prevention; Treatment adherence; Treatment for Prevention
MeSH Terms: conditions — HIV Infections; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated Intervention (Experimental): Five small group + 2 individual counseling behavioral intervention to simultaneously address HIV transmission risk reduction and HIV treatment adherence in men and women living with HIV/AIDS.
  Interventions: Behavioral: In The Mix
- Comparison Group (Active Comparator): Five small group + 2 individual counseling session intervention that serves as an attention control group. Content included stress reduction, nutrition, and exercise for health improvement.
  Interventions: Behavioral: Information Support Group

INTERVENTIONS:
Behavioral: In The Mix — Five small group + 2 individual counseling intervention designed to addresses HIV transmission risk behavior and HIV treatment adherence in men and women living with HIV/AIDS.
  Arms: Integrated Intervention
Behavioral: Information Support Group — Five small group + 2 individual counseling session intervention that serves as an attention control group. Content included stress reduction, nutrition, and exercise for health improvement.
  Arms: Comparison Group

SUMMARY:
HIV prevention interventions are needed to assist people living with HIV/AIDS to adhere to their medications and not transmit the virus to others. This study is testing a behavioral intervention designed to address both medication adherence and risk reduction in people living with HIV/AIDS. It is hypothesized that the experimental behavioral intervention will show improved medication adherence and safer sexual behaviors compared to a comparison group.

DETAILED DESCRIPTION:
Non-adherence to antiretroviral medications can lead to the development of treatment resistant genetic variants of HIV which can then be transmitted to sexual risk partners. Interventions are urgently needed to reduce the risk of HIV treatment resistance and the risks of transmitting HIV. This application proposes to test a theory-based behavioral intervention to simultaneously improve HIV treatment adherence and reduce HIV transmission risk behaviors in people living with HIV-AIDS. Grounded in behavioral theory, the experimental intervention will be delivered in a mixed format model with five group sessions preceded by and followed by one individual counseling session conducted by community-based group facilitators. The intervention will be conducted at an AIDS service organization in Atlanta. Men and women will be recruited from a variety of AIDS services and infectious disease clinics. Following informed consent and baseline assessments participants will be randomly assigned to receive either the (a) integrated HIV treatment adherence - risk reduction intervention or (b) a time-matched sexual risk reduction intervention, or (c) a time matched non-contaminating comparison intervention. Participants will be followed over the course of a 9-month observation period. Assessments will include measures of information, motivation, and behavioral skills pertaining to HIV treatment adherence and HIV transmission risks and risk reduction, medication adherence, sexual transmission risk behaviors, viral load, and CD4 cell counts. The study will test the hypothesis that a unified, integrated theory-based HIV treatment and risk reduction intervention will improve HIV treatment adherence, reduce HIV transmission risk behaviors, and improve health as indexed by viral load and CD4 cell counts. The study will also examine the influence of theoretical constructs on intervention outcomes. The intervention under investigation will be among the first to simultaneously address treatment adherence and risk behavior in an integrated model derived from a single, unified theory of health behavior. If shown effective, the intervention model will be ready for immediate dissemination to community services for people living with HIV-AIDS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older,
* Tested HIV positive,
* Able to provide informed consent.

Exclusion Criteria:

* Significant cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2005-03; Primary Completion 2009-10 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Computerized Interview or Sexual Transmission Risk Behavior | Baseline, 3, 6 and 9 months
Unannounced Phone Based Pill Counts for Medication Adherence | Baseline, 3, 6, 9 months

SECONDARY OUTCOMES:
Infectiousness Beliefs | Baseline, 3, 6, and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Seth C Kalichman, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Southeast HIV/AIDS Research and Evaluation Project, Atlanta, Georgia, United States